CLINICAL TRIAL: NCT02690194
Title: A Prospective Study Investigating the Use of Relaxation Prior to Medical Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Gianmichel Corrado, Gianmichel D. Corrado, MD, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00016464
Record Dates: First submitted 2016-02-09; First posted 2016-02-24 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Pain; Anxiety
Keywords: Buddhify; Stress; Anxiety; Relaxation Technique
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo Group (Placebo Comparator): 1. Pre-Placebo therapy
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  2. PLACEBO THERAPY SESSION
  3. Post-Placebo therapy/Pre-procedure
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  4. PROCEDURE
  5. Post-procedure -Rate pain level of procedure
  Interventions: Device: Placebo Group
- Experimental (Buddhify) Group (Experimental): 1. Pre-Buddhify therapy
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  2. BUDDHIFY THERAPY SESSION
  3. Post-Buddhify therapy/Pre-procedure
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  4. PROCEDURE
  5. Post-procedure -Rate pain level of procedure
  Interventions: Device: Buddhify Therapy
- Control Group (No Intervention): 1. Pre-Procedure
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  2. PROCEDURE
  3. Post-procedure -Rate pain level of procedure

INTERVENTIONS:
Device: Placebo Group — The placebo group will wear headphones and listen to nature sounds.
  Arms: Placebo Group
Device: Buddhify Therapy — The experimental group will complete a Buddhify relaxation therapy session, before their injection. This therapy consists of wearing headphones and listening to guided meditation instructions.
  Arms: Experimental (Buddhify) Group

SUMMARY:
The primary aim is to investigate the efficacy of Buddhify relaxation therapy in reducing the stress and anxiety levels of patients. The secondary aim is to investigate the effect of prior stress and anxiety levels on the perceived pain level of undergoing a medical procedure, reported post-procedure.

DETAILED DESCRIPTION:
Undergoing medical procedures is reported to cause stress and anxiety among many individuals.This can trigger the sympathetic nervous response, including decreased skin temperature, increased pulse, and increased blood pressure. While evolutionary advantageous, this response has deleterious effects on the healing process. Heightened stress levels can also trigger an increased release of cortisol, a naturally produced steroid hormone known to hinder the immune response. In response to high levels of stress, a patient's tolerance for pain decreases and the perceived pain level increases.

Relaxation techniques can assist in reducing the stress and anxiety levels of a patient, which allows for lower perceived pain and more rapid healing. Many relaxation techniques exist, including acupuncture, child life intervention, breathing therapy and guided imagery. Buddhify, a mobile application, incorporates breathing therapy and audio-guided imagery into brief relaxation sessions, with the goal of reducing the stress and anxiety levels of the user. This application presents a convenient option for patients to use prior to undergoing a procedure. If proven to be effective, this application could be more widely used to help reduce the stress level, anxiety level and subsequent perceived pain level of patients, ultimately improving their healing reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 14 and older undergoing an invasive procedure by Dr. Gianmichel Corrado at the Division of Sports Medicine of Boston Children's Hospital.

Exclusion Criteria:

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianmichel Corrado, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital - Sports Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae H, Bae H, Min BI, Cho S. Efficacy of acupuncture in reducing preoperative anxiety: a meta-analysis. Evid Based Complement Alternat Med. 2014;2014:850367. doi: 10.1155/2014/850367. Epub 2014 Sep 2. PMID 25254059
- [Background] Ko YL, Lin PC. The effect of using a relaxation tape on pulse, respiration, blood pressure and anxiety levels of surgical patients. J Clin Nurs. 2012 Mar;21(5-6):689-97. doi: 10.1111/j.1365-2702.2011.03818.x. Epub 2011 Nov 17. PMID 22092955
- [Background] Ebrecht M, Hextall J, Kirtley LG, Taylor A, Dyson M, Weinman J. Perceived stress and cortisol levels predict speed of wound healing in healthy male adults. Psychoneuroendocrinology. 2004 Jul;29(6):798-809. doi: 10.1016/S0306-4530(03)00144-6. PMID 15110929
- [Background] Worley CA. 'Why won't this wound heal?' Factors affecting wound repair. Dermatol Nurs. 2004 Aug;16(4):360-1. No abstract available. PMID 15471050
- [Background] Lim YC, Yobas P, Chen HC. Efficacy of relaxation intervention on pain, self-efficacy, and stress-related variables in patients following total knee replacement surgery. Pain Manag Nurs. 2014 Dec;15(4):888-96. doi: 10.1016/j.pmn.2014.02.001. Epub 2014 Jun 21. PMID 24957817
- [Background] Kiecolt-Glaser JK, Marucha PT, Malarkey WB, Mercado AM, Glaser R. Slowing of wound healing by psychological stress. Lancet. 1995 Nov 4;346(8984):1194-6. doi: 10.1016/s0140-6736(95)92899-5. PMID 7475659
- [Background] Heilbrunn BR, Wittern RE, Lee JB, Pham PK, Hamilton AH, Nager AL. Reducing anxiety in the pediatric emergency department: a comparative trial. J Emerg Med. 2014 Dec;47(6):623-31. doi: 10.1016/j.jemermed.2014.06.052. Epub 2014 Sep 27. PMID 25271180
- [Derived] Sugimoto D, Slick NR, Mendel DL, Stein CJ, Pluhar E, Fraser JL, Meehan WP 3rd, Corrado GD. Meditation Monologue can Reduce Clinical Injection-Related Anxiety: Randomized Controlled Trial. J Evid Based Integr Med. 2021 Jan-Dec;26:2515690X211006031. doi: 10.1177/2515690X211006031. PMID 33904781

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Control group data was not analyzed for all measures
Groups:
- Placebo Group: 1. Pre-Placebo therapy
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  2. PLACEBO THERAPY SESSION
  3. Post-Placebo therapy/Pre-procedure
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  4. PROCEDURE
  5. Post-procedure -Rate pain level of procedure
  Placebo Group: The placebo group will wear headphones and listen to nature sounds.
- Experimental (Buddhify) Group: 1. Pre-Buddhify therapy
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  2. BUDDHIFY THERAPY SESSION
  3. Post-Buddhify therapy/Pre-procedure
     * Blood pressure, pulse, and respiration rate
     * State-Trait Anxiety Inventory
  4. PROCEDURE
  5. Post-procedure -Rate pain level of procedure
  Buddhify Therapy: The experimental group will complete a Buddhify relaxation therapy session, before their injection. This therapy consists of wearing headphones and listening to guided meditation instructions.
Period: Overall Study
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Started | 17 | 18 | 19
Completed | 16 | 14 | 19
Not Completed | 1 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: For the control group there were no post-therapy/pre-procedure data collected because there was no therapy for the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group | Total
Number analyzed (Participants) | 16 | 14 | 19 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 2 | 5
  Between 18 and 65 years | 11 | 8 | 10 | 29
  >=65 years | 3 | 5 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (18.0) | 53.9 (15.8) | 55.5 (17.1) | 52.4 (2.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 14 | 35
  Male | 6 | 3 | 5 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pre-therapy/Pre-procedure Stress Level Measured by Blood Pressure
Description: Pre-therapy/pre-procedure stress level measured by blood pressure in mmHg
Time Frame: Pre-therapy/pre-procedure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
mmHg
  BP-Systolic | 121.9 (17.5) | 121.9 (9.5) | 127.3 (14.1)
  BP-Diastolic | 77.2 (10.8) | 78.9 (8.1) | 82.2 (11.3)

2. Primary Outcome: Pre-therapy/Pre-procedure Stress Level Measured by Pulse
Description: Pre-therapy/pre-procedure stress level measured by pulse in beats per minute.
Time Frame: Pre-therapy/pre-procedure
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
Beats per minute | 75.6 (14.3) | 66.4 (14.4) | 69.5 (11.2)

3. Primary Outcome: Pre-therapy/Pre-procedure Stress Level Measured by Respiratory Rate
Description: Pre-therapy/pre-procedure stress level measured by respiratory rate in breaths per minute.
Time Frame: Pre-therapy/pre-procedure
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
Breaths per minute | 16.1 (3.0) | 14.0 (2.1) | 14.4 (2.1)

4. Primary Outcome: Pre-therapy/Pre-procedure Anxiety Level
Description: Pre-therapy/pre-procedure anxiety level measure by the State-Trait Anxiety Inventory. The scale ranges from a minimum score of 40 to a maximum score of 160 with a higher score indicating higher levels of anxiety.
Time Frame: Pre-therapy/pre-procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
score on a scale
  S-Anxiety Score | 33.1 (7.2) | 34.4 (10.9) | 31.4 (7.1)
  T-Anxiety Score | 35.6 (6.1) | 34.0 (7.6) | 32.4 (9.4)

5. Secondary Outcome: Post-therapy/Pre-procedure Change in Stress Level Measured by Pulse
Description: Post-therapy/pre-procedure change in stress level measured by pulse in beats per minute. Value at prost-therapy/pre-procedure minus value at pre-therapy/pre-procedure.
Time Frame: Post-therapy/pre-procedure
Population: No data were collected for the control group in this Outcome Measure
Measure: Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Placebo Group | Experimental (Buddhify) Group
Number analyzed (Participants) | 16 | 14
Beats per minute | -0.11 [-8.1 to 7.8] | 3.48 [-5.1 to 12.1]

6. Secondary Outcome: Post-therapy/Pre-procedure Change in Stress Level Measured by Respiration Rate
Description: Post-therapy/pre-procedure stress level measured by respiratory rate in breaths per minute. Value at post-therapy/pre-procedure minus value at pre-therapy/pre-procedure.
Time Frame: Post-therapy/pre-procedure
Population: No data were collected for the control group in this Outcome Measure.
Measure: Mean (95% Confidence Interval); unit: Breaths per minute
Arm/Group | Placebo Group | Experimental (Buddhify) Group
Number analyzed (Participants) | 16 | 14
Breaths per minute | -0.14 [-0.78 to 0.51] | -0.70 [-1.4 to 0.0]

7. Secondary Outcome: Post-therapy/Pre-procedure Change in Anxiety Level
Description: Post-therapy/Pre-procedure change in anxiety level measure by the State-Trait Anxiety Inventory. Value at post-therapy/pre-procedure minus value at pre-therapy/pre-procedure. The scale ranges from a minimum score of 40 to a maximum score of 160 with a higher score indicating higher levels of anxiety.
Time Frame: Post-therapy/pre-procedure
Population: No data were collected for the control group in this Outcome Measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Experimental (Buddhify) Group
Number analyzed (Participants) | 16 | 14
score on a scale
  S-Anxiety Score | -2.82 [-8.4 to 2.7] | -12.3 [-18.3 to -6.3]
  T-Anxiety Score | -8.44 [-15.2 to -1.7] | -3.92 [-11.2 to 3.4]

8. Secondary Outcome: Post-therapy/Pre-procedure Change in Stress Level Measured by Blood Pressure
Description: Post-therapy/pre-procedure change in stress level measured by blood pressure measured in mmHg. Value at post-therapy/pre-procedure minus value at pre-therapy/pre-procedure.
Time Frame: Post-therapy/Pre-procedure
Population: No data were collected for the control group in this Outcome Measure.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo Group | Experimental (Buddhify) Group
Number analyzed (Participants) | 16 | 14
mmHg
  BP-Systolic | 3.9 [-3.5 to 11.3] | -1.1 [-9.1 to 6.9]
  BP-Diastolic | 7.0 [1.5 to 12.4] | -1.2 [-7.1 to 4.7]

9. Secondary Outcome: Perceived Pain Level of the Procedure as Assessed by the Wong-Baker FACES Pain Rating Scale
Description: Perceived pain level of the procedure as assessed by the Wong-Baker FACES pain rating scale 1-10. A score of 1 indicates "no hurt" (a better outcome) while a score of 10 indicates "hurts worst" (worst outcome).
Time Frame: Immediately post-procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
score on a scale | 1.5 (1.6) | 1.9 (1.9) | 1.4 (1.5)

10. Secondary Outcome: Drink in Last Hour
Description: Indication of if the patient has had a drink in the last hour
Time Frame: Pre-therapy/Pre-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
Participants
  No | 8 | 4 | 11
  Yes | 8 | 10 | 8

11. Secondary Outcome: Eat in Last Hour
Description: Indication of if the patient has eaten in the last hour
Time Frame: Pre-therapy/Pre-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
Participants
  No | 13 | 11 | 12
  Yes | 3 | 3 | 7

12. Secondary Outcome: Exercise in Last Hour
Description: Indication of if the patient has exercised in the last hour
Time Frame: Pre-therapy/Pre-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
Participants
  No | 16 | 9 | 17
  Yes | 0 | 5 | 2

13. Secondary Outcome: Injection Experiences
Description: Indication of prior injection experiences
Time Frame: Pre-therapy/Pre-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 16 | 14 | 19
Participants
  No | 5 | 5 | 6
  Yes | 10 | 9 | 13
  Data Not Collected | 1 | 0 | 0

14. Secondary Outcome: Number of Injections
Description: Average number of injections for patients that indicated that they previously have had injections
Time Frame: Pre-therapy/Pre-procedure
Population: Patients that have had injections in the past
Measure: Mean (Standard Deviation); unit: Number of injections
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
Number analyzed (Participants) | 10 | 9 | 19
Number of injections | 5.8 (8.9) | 5.2 (3.4) | 4.3 (2.6)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Placebo Group | Experimental (Buddhify) Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes